CLINICAL TRIAL: NCT07064551
Title: Evaluation Study of Medical-Social Collaboration Model for Middle-aged and Older Adults With Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority Hong Kong West Cluster (Unknown); Hospital Authority Hong Kong East Cluster (Unknown); Hospital Authority Kolwoon Central Cluster (Unknown)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-649
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Depressive symptoms; Mental health; Medical-social collaboration; Integrated health and social care; Stepped-care intervention
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Masking Description: Masking was no possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JC JoyAge stepped-care model (Experimental)
  Interventions: Behavioral: Cognitive behavioural therapy-based stepped-care intervention; Other: Self-management booklet
- Usual care with minimal support (Other)
  Interventions: Other: Self-management booklet

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy-based stepped-care intervention — After initial clinical assessment, participants will be offered interventions based on their depressive symptom severity (Patient Health Questionnaire-9-item [PHQ-9]). Mild symptoms (PHQ-9=5-9): 6 weekly low intensity CBT-based group intervention sessions led by trained clinical social workers, with 2 booster sessions as necessary. Moderate symptoms (PHQ-9=10-14): 6 weekly high intensity CBT-based group intervention sessions led by trained clinical social workers, with 2 booster sessions as necessary. Moderately severe symptoms (PHQ-9≥15): high intensity individual or group CBT-based intervention. Trained peer supporters will be matched to participants to walk them through the process with regular follow-up.
  Arms: JC JoyAge stepped-care model
Other: Self-management booklet — The booklet incorporates components of behavioural activation, which encourages participants to engage in meaningful activities in daily life to change their mood. Trained research assistants will regularly check in with the participants to monitor their depressive symptoms.

SUMMARY:
The goal of this clinical trial is to learn if a medical-social collaboration model works to reduce depressive symptoms in middle-aged and older adults with subsyndromal depressive symptoms who are waiting for their first psychiatric appointment. Secondary outcomes of the study include reduced anxiety symptoms, reduced loneliness, reduced rumination, reduced self-criticism, improved self-reassurance, improved resilience, improved self-efficacy, improved health-related quality of life, as well as improved quality-adjusted life years, and reduced healthcare service utilisation.

Researchers will compare a medical-social collaboration model to a self-management booklet.

Participants will:

* Receive CBT-based stepped-care interventions through the medical-social collaboration model or a self-management booklet.
* Complete a survey about their mental health and service use every three months until their first psychiatric appointment.

ELIGIBILITY:
Inclusion Criteria:

* Currently awaiting psychiatric services provided by the Hospital Authority
* Have depressive symptoms of at least mild severity
* Able to provide informed consent

Exclusion Criteria:

* A known history of autism spectrum disorder, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia
* Imminent suicidal risk (temporary exclusion)
* Communication difficulties that preclude participation

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Depressive Symptoms | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Patient Health Questionnaire-9 (PHQ-9); range 0-27; higher scores indicate higher levels of depressive symptoms (worse outcome)

SECONDARY OUTCOMES:
Changes in Anxiety Symptoms | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Generalized Anxiety Disorder 2-item scale (GAD-2); range 0-6; higher scores indicate higher levels of anxiety symptoms (worse outcome)
Changes in Loneliness | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  UCLA Loneliness Scale (UCLA-3); range 0-9; higher scores indicate higher levels of perceived loneliness (worse outcome)
Changes in Health Service Use | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Self-reported use of mental health services and medication in the past three months.
  Service data from Hospital Authority, covering information on outpatient visits, hospitalisation days, Accident and Emergency service utilisation, types of medications and operations, and any other major cost items that may be affected by depression with cost implications.
Changes in Health-Related Quality of Life | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  EQ-5D-5L; range 0-1; higher scores indicate higher levels of health-related quality of life (better outcome)

OTHER OUTCOMES:
Self-Criticism and Self-Reassurance | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Short Form of Forms of Self-Criticizing/Attacking and Self-Reassuring Scale (FSCRS-SF); higher scores indicate a greater sense of inadequacy (score 0-20) (worse outcome), self-hate (score 0-16) (worse outcome), and self-reassurance (score 0-20) (better outcome)
Rumination | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Ruminative Response Scale - Brooding Subscale (RRS-Brooding); range 0-15; higher scores indicate higher frequency of depressive rumination (worse outcome)
Resilience | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Connor-Davidson Resilience Scale 2-Item (CD-RISC-2); range 0-8; higher scores indicate higher levels of resilience or better equipped to bounce back after stressful events (better outcome)
General Self-Efficacy | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Single-item General Self-Efficacy Scale (SI-DSES); range 1-5; higher scores indicate higher levels of self-efficacy (better outcome)
Stressful Events | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Self-reported stressful events, e.g. illness, death of close relative/friends.
Perceived Neighbourhood Environment | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months
  Self-perceived convenience to access leisure, shopping, and community facilities and social and medical services

CONTACTS AND LOCATIONS:
Overall Officials: Terry YS Lum, PhD, Principal Investigator — The University of Hong Kong; Gloria HY Wong, PhD, Principal Investigator — University of Reading; Wai Chi Chan, MBChB, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to participant confidentiality reasons.